CLINICAL TRIAL: NCT06725004
Title: Oxytocin Versus Human Chorionic Gonadotropin as Trigger in Ovulation Induction Cycles: A Randomized Controlled Trial
Brief Title: Oxytocin Versus Human Chorionic Gonadotropin as Trigger in Ovulation Induction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shakeela Ishrat (Other)
Responsible Party: Sponsor-Investigator, Shakeela Ishrat, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Organization: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4221
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-05

CONDITIONS: Ovulation Induction; Polycystic Ovary Syndrome
Keywords: Ovulation induction; Polycystic Ovary Syndrome; Oxytocin; Human Chorionic Gonadotropin (HCG)
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Oxytocin; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): Participants will receive injection oxytocin 10 mg intramuscular as trigger for ovulation induction
  Interventions: Drug: Oxytocin
- Human Chorionic Gonadotropin (Active Comparator): Participants will receive injection Human Chorionic Gonadotropin 5000 IU intramuscular as trigger for ovulation induction
  Interventions: Drug: Human Chorionic Gonadotropin

INTERVENTIONS:
Drug: Oxytocin — Injection Oxytocin 10 mg intramuscular as trigger for ovulation induction
  Arms: Oxytocin
Drug: Human Chorionic Gonadotropin — Injection Human Chorionic Gonadotropin 5000 IU intramuscular as trigger for ovulation induction
  Arms: Human Chorionic Gonadotropin

SUMMARY:
The goal of this clinical trial is to learn if injection oxytocin can be used as trigger in ovulation induction cycles in infertile women with polycystic ovary syndrome. The main questions it aims to answer are:

* Does injection oxytocin have similar ovulation rate as injection human chorionic gonadotropin (hCG) when used as trigger?
* Does injection oxytocin have similar pregnancy rate as injection human chorionic gonadotropin (hCG) when used as trigger?

Researchers will compare injection oxytocin to injection hCG to see if injection oxytocin is as effective as injection hCG as trigger in ovulation induction cycles in infertile women with polycystic ovary syndrome.

Participants will

* Take injection oxytocin or injection hCG as trigger over three subsequent ovulation induction cycles
* Be checked for ovulation by follicular rupture in TVS after 36 hours or raised serum progesterone level on day 7 after trigger
* Be checked for pregnancy by urine pregnancy test kit after missed period

DETAILED DESCRIPTION:
This is an open label randomized controlled trial. After baseline transvaginal sonography (TVS), all the participants will be given tablet letrozole 5 mg or more from day 2 to day 6 of their menstrual cycle. Then participants will be followed up by TVS for follicular maturation and endometrial thickness.When the size of mature follicle will be at least 18mm , then participants will be randomized into experimental group and comparator group. The participants in experimental group will receive inj. (injection) oxytocin 10 IU (Inj. Linda 10 unit, Nuvista Pharmaceuticals Limited) intramuscular as trigger and the participants in control group received Inj. hCG 5000 IU (Inj. hCG 5000 IU, Popular Pharmaceuticals Limited) intramuscular as trigger. Participants will be followed up 36 hours after injection by TVS for follicular rupture. On the 7th day following oxytocin or hCG injection, serum progesterone level will be measured by chemiluminescent immunoassay . Participants will be followed until the next cycle for conception. If conception does not occur, then the procedure will be repeated in next cycle for 3 cycles.

Random sequence generation will be done by computer generated random numbers after permuted block randomization. Allocation concealment will be done by serially numbered closed envelops. Each envelop will be labeled with a serial number and has a card inside noting the intervention drug. A sample size of 24 in each group will be calculated to detect a non-inferiority margin difference between the group proportions with 80.9% power and the level of significance 0.05. Considering 10% patients drop out, 30 participants will be recruited in each group.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women with polycystic ovary syndrome
* Age less than 40 years
* Had ovulation induction with letrozole, with at least one mature follicle detected on folliculometry

Exclusion Criteria:

* Male factor abnormality
* Bilateral tubal block
* Any pelvic pathology like pelvic inflammatory diseases
* Any uterine abnormality
* Ovarian cysts
* Any cardiovascular diseases or other systemic diseases
* Hyperprolactinemia or thyroid dysfunction
* Any drugs that affect the functions of hypothalamus, pituitary gland, and gonads
* Any known hypersensitivity to oxytocin

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants having ovulation | 1 week
  Number of participants having ovulation defined by findings on TVS after 36 hours and/or serum progesterone level 7th day after triggering

SECONDARY OUTCOMES:
Number of participants having pregnancy | 3 weeks
  Number of participants having pregnancy determined by urinary pregnancy kit test after missed period.

CONTACTS AND LOCATIONS:
Overall Officials: Shakeela Ishrat, FCPS,MS, Study Director — Bangladesh Medical University
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehrotra S, Singh U, Gupta HP, Tandon I, Saxena P. A prospective double blind study comparing the effects of oxytocin and human chorionic gonadotrophin as trigger for ovulation. J Obstet Gynaecol. 2014 Jan;34(1):13-6. doi: 10.3109/01443615.2013.822479. PMID 24359041
- [Background] George K, Kamath MS, Nair R, Tharyan P. Ovulation triggers in anovulatory women undergoing ovulation induction. Cochrane Database Syst Rev. 2014 Jan 31;2014(1):CD006900. doi: 10.1002/14651858.CD006900.pub3. PMID 24482059